CLINICAL TRIAL: NCT05914077
Title: Aspiration of Duodenopancreatic Juice After Secretin Stimulation (ADPJ-secr-) vs Endoscopic Aspiration (EUS-FNA) for Molecular Analysis of Intraductal Papillary Mucinous Intraductal Neoplasia (IPMN).
Brief Title: Aspiration of Duodenopancreatic Juice After Secretin Stimulation vs Endoscopic Aspiration for Molecular Analysis of Intraductal Papillary Mucinous Intraductal Neoplasia.
Acronym: RESCUE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-002764-79
Record Dates: First submitted 2023-05-04; First posted 2023-06-22 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Intraductal Papillary Mucinous Neoplasm of Pancreas
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms | interventions — Secretin; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Duodenopancreatic aspiration after secretin stimulation + EUS-FNA (Experimental): Duodenopancreatic aspiration after secretin stimulation will be performed followed by endoscopic ultrasound-guided fine needle aspiration (EUS-FNA)
  Interventions: Drug: Secretin; Procedure: Endoscopic aspiration; Procedure: Endoscopic ultrasound-guided fine needle aspiration
- EUS-FNA + duodenopancreatic aspiration after secretin stimulation (Experimental): Endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) will be performed followed by duodenopancreatic aspiration after secretin stimulation
  Interventions: Drug: Secretin; Procedure: Endoscopic aspiration; Procedure: Endoscopic ultrasound-guided fine needle aspiration

INTERVENTIONS:
Drug: Secretin — Secretin will be administered intravenous during 1 minute at a dose of 0,2 μg/Kg previous to the endoscopic procedure.
Procedure: Endoscopic aspiration — Endoscopic aspiration of duodenopancreatic juice after secretin stimulation
Procedure: Endoscopic ultrasound-guided fine needle aspiration — Endoscopic ultrasound-guided fine needle aspiration of intraductal papillary mucinous intraductal neoplasia (IPMN).

SUMMARY:
Study to evaluate aspiration of duodenopancreatic juice after secretin stimulation (ADPJ-secr)versus endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) for molecular analysis of intraductal papillary mucinous intraductal neoplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Be a man or woman over 18 years of age.
2. Willing to comply with the study procedures described in the protocol.
3. Willing and able to give written informed consent.
4. Meet at least one of the following three criteria in relation to the diagnosis or prognosis of IPMN:

   4.1 Diagnosis of IMPN based on evidence of major criteria or existence of at least 2 minor criteria. Major criterion: Typical findings on MRI and/or EUS (single or multiple cysts with clear ductal communication and/or focal or diffuse dilatation # 5 mm in diameter of the main pancreatic duct without apparent obstructive cause). Minor criteria: a) Mucosecretory cells and/or extracellular mucin on cytological examination of intracystic fluid. b) Clear mucoid or filmy appearance of the intracystic fluid. c) Intracystic fluid CEA concentration >192 ng/mL or intracystic glucose < 50 mg/dL.

   4.2 IPMN with cysts with a diameter # 10 mm and/or focal or diffuse dilatation of the main pancreatic duct with a diameter # 7 mm requiring EUS-FNA for diagnostic purposes or to assess risk or existence of malignancy following the main clinical practice guidelines.

   4.3 IPMN with indication for surgical resection of the lesion.
5. In case of a woman of childbearing age*, willing to use highly effective contraception or practice sexual abstinence from the screening visit until one week after undergoing the procedure under study. Highly effective contraceptive methods will include: combined oral, intravaginal or transdermal hormonal contraceptives (containing oestrogens and progestogens) associated with ovulation inhibition; oral, injectable or implantable progestogen-only hormonal contraception associated with ovulation inhibition; intrauterine device; intrauterine hormone-releasing system; bilateral tubal occlusion; vasectomised partner; and sexual abstinence. 6. If you are a woman of childbearing age, be willing to undergo a urine pregnancy test prior to inclusion in the study.

Exclusion Criteria:

1. History of surgery that prevents endoscopic access to the major duodenal papilla in the case of ADPJ-secr, or to the area of the stomach or intestine from which to perform FNA.
2. History of acute pancreatitis during the 30 days prior to inclusion.
3. Pregnant women, women who may become pregnant during the month prior to inclusion or women who are breastfeeding.
4. Coagulopathy (PT < 25%, INR > 1.5, platelets < 50,000/mL) preventing FNA.
5. Renal failure with GFR < 30 mL/min or patients on dialysis.
6. Known hypersensitivity to any component of the ChiRhoStim® (human secretin) formulation.
7. Any clinically relevant medical condition that, in the opinion of the investigator, makes the patient unfit to participate in the study (underlying haematological disorders, autoimmune disease, immunodeficiency, gastrointestinal, psychiatric, renal, hepatic and cardiopulmonary disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with IPMN with GNAS and KRAS mutations in intracystic fluid obtained by EUS-FNA versus pancreatic juice obtained by ADPJ-secr after both techniques. | Through study completion, an average of 30 months
  In intracystic fluid obtained by EUS-FNA versus pancreatic juice obtained by ADPJ-secr after both techniques.

SECONDARY OUTCOMES:
Proportion of patients with IPMN with Tp53 mutations. | Through study completion, an average of 30 months
  In samples obtained by EUS-FNA versus ADPJ-secr after performing both techniques, in the subgroup of patients undergoing pancreatic resection within 12 months after study entry.
DNA concentration expressed in ng/µl | Through study completion, an average of 30 months
  In samples obtained by EUS-FNA versus ADPJ-secr after performing both techniques.
Proportion of suitable samples obtained by the two techniques under study (ADPJ-secr and EUS-FNA) for molecular analysis. | Through study completion, an average of 30 months
  A sample is defined as suitable when it is read by the Qubit fluorometer, which only detects full double-stranded DNA suitable for molecular analysis.
Proportion of patients undergoing pancreatic resection with a pathological diagnosis of IPMN who have mutations in GNAS and/or KRAS | Through study completion, an average of 30 months
  In samples obtained by EUS-FNA versus ADPJ-secr within 12 months of study entry.
Proportion of patients undergoing pancreatic resection without a pathological diagnosis of IPMN who do not have GNAS and/or KRAS mutations | Through study completion, an average of 30 months
  In samples obtained by EUS-FNA versus ADPJ-secr within 12 months of study entry.
Proportion of patients undergoing pancreatic resection with Tp53 mutations | Through study completion, an average of 30 months
  In samples obtained by both techniques under study (ADPJ-secr vs EUS-FNA) who have advanced neoplasia in the surgical resection specimen after surgery performed within 12 months after study inclusion.
  Advanced neoplasia is defined as the presence of IPMN with high-grade dysplasia or IMPN with associated invasive carcinoma according to Lokuhetty D, et al. Digestive SystemTumours: WHO Classification of Tumours, International Agency for Research on Cancer, 2019.
Proportion of patients undergoing pancreatic resection without Tp53 mutations. | Through study completion, an average of 30 months
  In samples obtained by both techniques under study (ADPJ-secr vs EUS-FNA) who do not have advanced neoplasia in the surgical resection specimen after surgery performed within 12 months after inclusion in the study.
  Advanced neoplasia is defined as the presence of IPMN with high-grade dysplasia or IPMN with associated invasive carcinoma according to Lokuhetty D, et al. Digestive System Tumours: WHO Classification of Tumours, International Agency for Research on Cancer, 2019.
To evaluate association between mutational status in the samples obtained by both techniques in relation to morphological characteristics of the lesion (diameter of the largest cystic lesion) obtained by EUS. | Through study completion, an average of 30 months
  To compare if diameter of the largest cystic lesion in mm is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status in the samples obtained by both techniques in relation to morphological characteristics of the lesion (maximum diameter of the main pancreatic duct) obtained by EUS. | Through study completion, an average of 30 months
  To compare if median maximum diameter of the main pancreatic duct assessed by EUS and measured in mm is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status in the samples obtained by both techniques in relation to morphological characteristics of the lesion (type of main pancreatic duct dilatation) obtained by EUS. | Through study completion, an average of 30 months
  To compare if the proportion of patients that present a segmental main pancreatic duct dilatation assessed by EUS is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status in the samples obtained by both techniques in relation to morphological characteristics of the lesion (location of the lesion) obtained by EUS. | Through study completion, an average of 30 months
  To compare if the proportion of cystic lesions located in the pancreatic head, pancreatic body or pancreatic tail assessed by EUS are different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status in the samples obtained by both techniques in relation to morphological characteristics of the lesion (presence > 1 cystic lesion) obtained by EUS. | Through study completion, an average of 30 months
  To compare if the proportion of patients with > 1 pancreatic cystic lesion assessed by EUS is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status in the samples obtained by both techniques in relation to morphological characteristics of the lesion (mural nodules) obtained by EUS. | Through study completion, an average of 30 months
  To compare if the proportion of patients that present mural nodules assessed by EUS is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status in the samples obtained by both techniques in relation to morphological characteristics of the lesion (signs of chronic pancreatitis) obtained by EUS. | Through study completion, an average of 30 months
  To compare if the proportion of patients that present features of chronic pancreatitis assessed by EUS is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status in the samples obtained by both techniques in relation to morphological characteristics of the lesion (intraductal calcifications) obtained by EUS. | Through study completion, an average of 30 months
  To compare if the proportion of patients that present intraductal calcifications assessed by EUS is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status in the samples obtained by both techniques in relation to morphological characteristics of the lesion (pancreatic atrophy) obtained by EUS. | Through study completion, an average of 30 months
  To compare if the proportion of patients that present pancreatic atrophy assessed by EUS is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to age | Through study completion, an average of 30 months
  To compare if median of age measured in years is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to sex | Through study completion, an average of 30 months
  To compare if the proportion of male or female patients are different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to smoking | Through study completion, an average of 30 months
  To compare if the proportion of patients with reported active smoking is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to chronic alcohol consumption | Through study completion, an average of 30 months
  To compare if the proportion of patients with high risk chronic alcohol consumption (> 21 standard drinks for men, > 14 standard drinks for women) is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to hypertension | Through study completion, an average of 30 months
  To compare if the proportion of patients with hypertension is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to type 2 diabetes mellitus | Through study completion, an average of 30 months
  To compare if the proportion of patients with type 2 diabetes mellitus is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to heart failure | Through study completion, an average of 30 months
  To compare if the proportion of patients with chronic heart failure is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to chronic liver disease. | Through study completion, an average of 30 months
  To compare if the proportion of patients with chronic liver disease is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to chronic kidney disease. | Through study completion, an average of 30 months
  To compare if the proportion of patients with chronic kidney disease is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to neoplasms. | Through study completion, an average of 30 months
  To compare if the proportion of patients with previous neoplasm in past medical history is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to history of acute pancreatitis | Through study completion, an average of 30 months
  To compare if the proportion of patients with history of acute pancreatitis in past medical history is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to previous diagnosis of chronic pancreatitis | Through study completion, an average of 30 months
  To compare if the proportion of patients with history of chronic pancreatitis in past medical history is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to family history (1st degree) of pancreatic cancer | Through study completion, an average of 30 months
  To compare if the proportion of patients with history of pancreatic cancer in first degree relatives is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to time since diagnosis of IPMN | Through study completion, an average of 30 months
  To compare if time since diagnosis of IPMN measured in years is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to morphological type of IPMN | Through study completion, an average of 30 months
  To compare if the proportions of patients with MD-IPMN, BD-IPMN or mixed-type IPMN are different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of amylase | Through study completion, an average of 30 months
  To compare if mean blood levels of amylase measured in U/L is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of lipase | Through study completion, an average of 30 months
  To compare if mean blood levels of lipase measured in U/L is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of creatinine | Through study completion, an average of 30 months
  To compare if mean blood levels of creatinine measured in mg/dl is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of total bilirrubin | Through study completion, an average of 30 months
  To compare if mean blood levels of total bilurrubin measured in mg/dl is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of AST | Through study completion, an average of 30 months
  To compare if mean blood levels of AST measured in U/L is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of ALT (U/L) | Through study completion, an average of 30 months
  To compare if mean blood levels of ALT measured in U/L is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of GGT (U/L) | Through study completion, an average of 30 months
  To compare if mean blood levels of GGT measured in U/L is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of alkaline phosphatase (U/L) | Through study completion, an average of 30 months
  To compare if mean blood levels of alkaline phosphatase measured in U/L is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of hemoglobin (g/L) | Through study completion, an average of 30 months
  To compare if mean blood levels of hemoglobin measured in g/l is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of platelets (U/L) | Through study completion, an average of 30 months
  To compare if mean blood total count of platelets measured in units per microliter is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of CA 19.9 (u/L) | Through study completion, an average of 30 months
  To compare if mean blood levels of CA 19.9 measured in U/L is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of CEA (U/l) | Through study completion, an average of 30 months
  To compare if mean blood levels of CEA measured in U/L is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To evaluate association between mutational status (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]) in the samples obtained by both techniques under study (ADPJ-secr and EUS-FNA) in relation to blood levels of glycated hemoglobin.(%). | Through study completion, an average of 30 months
  To compare if mean blood levels of glycated hemoglobin measured in % is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]).
To assess whether mutational status predicts the occurrence of adverse effects associated with the techniques under study at 24 hours and 7 days following the performance of the techniques under study. | Through study completion, an average of 30 months
  To compare if the proportion of patients with adverse effects associated with the techniques under study at 24 hours and 7 days is different between both groups of study (mutated GNAS/KRAS versus non-mutated GNAS/KRAS [wild type]). Adverse effects will be reported following the American Society of Gastrointestinal Endoscopy (ASGE) (P.B. Cotton, et al. Gastrointest Endosc, 2010) and the WHO Toxicity Grading Scale for Determining the Severity of Adverse Events, 2003.
Proportion of patients with Serious Adverse Events | At 24 hours and 7 days after the techniques under study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain